CLINICAL TRIAL: NCT06355154
Title: Effects of Moderate Carbohydrate Consumption on Metabolic and Obstetric Outcomes in Pregnant Women With Insulin-treated Diabetes- A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 069823- HMO-CTIL
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes in Pregnancy
Keywords: Diabetes in pregnancy; Glycemic balance; Low Carbohydrates; Time in range; Ketosis
MeSH Terms: conditions — Diabetes, Gestational; Ketosis

STUDY DESIGN:
Intervention Model Description: Open label, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Standard of Care diet (No Intervention): (a diet that includes at least 175 grams of carbohydrates per day or more/ >40% CHO, SCD)
- The moderate carbohydrate diet (Experimental): (a diet with 120 grams of carbohydrates and customized according to pregnancy requirements/ <40% CHO, MCD)
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — The intervention will contain a diet with a reduced amount of carbohydrates compared to the standard treatment today but without caloric restriction.
  Arms: The moderate carbohydrate diet

SUMMARY:
Diabetes during pregnancy increases maternal and fetal complications, necessitating optimal glycemic control. The standard care diet (SCD, ≥175g/day carbohydrate) lacks robust evidence, particularly for pregnancies requiring intensive insulin treatment (IIT). This RCT investigates whether a moderate carbohydrate diet (MCD, ≤120g/day) versus SCD improves glycemic control and alters metabolomic profiles in pregnant individuals on IIT.

Aims: To compare the efficacy and safety of a SCD versus MCD on glycemic control, metabolomic signatures, and pregnancy outcomes in pregnant individuals on IIT.

DETAILED DESCRIPTION:
Effects of moderate carbohydrate consumption on metabolic and obstetric outcomes in pregnant women with insulin-treated diabetes- A randomized controlled trial

1. Scientific Background:

   1.1 Diabetes Mellitus in Pregnancy: Diabetes during pregnancy (pre-gestational type 1 or 2, or gestational diabetes) is associated with complications for both the mother (polyhydramnios, miscarriage, hypertension, preeclampsia, need for instrumental delivery) and the fetus/neonate (birth defects, macrosomia, shoulder dystocia, respiratory distress, hyperbilirubinemia, hypoglycemia). (1),(2) ,(3),(4). The incidence of all forms of diabetes during reproductive age is increasing(5).

   1.2 Dietary carbohydrate consumption during pregnancy: Current guidelines recommend a minimum carbohydrate consumption of 175g/day for all pregnant women, regardless of diabetes status. This is based on a theoretical calculations rather than clinical evidence (6). Some concerns with carbohydrate restriction during pregnancy include disrupting the maternal-fetal glucose gradient, increased fetal ketone exposure, micronutrient deficiency, and increased maternal triglycerides/free fatty acids(7).

   However, recent studies found no correlation between moderate carbohydrate restriction (<175g/day but >120g/day) and increased ketosis(8),(9),(10). Reducing carbohydrates may help reduce postprandial hyperglycemia in patients on intensive insulin therapy(11),(12).These findings call into question the hypothetical assumption that a minimum of 175 gr of CHO is required during pregnancy.
2. Research Objective:

   The primary objectives of the trial are to determine:
   * To assess the effectiveness and safety of moderate carbohydrate consumption restriction (MCD) in enhancing glycemic control.
   * To investigate the impact of MCD on the metabolomic profile of pregnant individuals with diabetes requiring intensive insulin treatment (MDI/CII).
3. Expected Significance:

The importance of this study lies in:

1. Challenging the commonly accepted but theoretical recommendation of 175g/day minimum carbohydrate intake during pregnancy.
2. Evaluating if moderate carbohydrate restriction can improve glycemic control and pregnancy outcomes in women with diabetes requiring intensive insulin therapy, without major adverse effects.

4.Detailed Description of the Proposed Research: 4.1 Study Design: This is an open label, randomized controlled trial comprising 120 pregnant individuals (18-45 years) with any form of diabetes requiring intensive insulin therapy. Pregnant individuals on IIT will be randomized to standard carbohydrate diet (>175g/day) or moderate carbohydrate diet (120g/day) group.

Key Measurements/Data Collection:

* Continuous glucose monitoring (CGM) to assess time in range (TIR) and other glycemic parameters.
* Anthropometrics (weight, height, BMI).
* Dietary intake data (FFQs, 24-hr recalls, 3-day food diaries).
* Blood tests (HbA1c, glucose, c-peptide, lipids, etc).
* Fetal growth monitoring via ultrasound.
* Cord blood c-peptide at delivery.
* Neonatal and maternal post-delivery outcomes (mode of delivery, weight, complications, etc).
* Maternal metabolomics (fasting blood sample). 4.3 Study Visits:
* Screening/baseline visit to assess eligibility.
* Dietary counseling and medical team visits every 2 weeks until 32 weeks, then weekly or as be decided by the medical team according to patients needs.
* Fetal ultrasounds start at 28 weeks, twice monthly or more.
* Final visit at 35-38 weeks for metabolomics sample. 4.4 Safety Monitoring:
* No intended calorie restriction.
* CGM to adjust insulin and avoid hypoglycemia.
* Home ketone monitoring.
* Ultrasound fetal growth monitoring. 4.5 Metabolomics Analysis:
* LC-MS analysis to detect >400 metabolites.
* Assess effects on micronutrients, carbs, lipids, ketones, amino acids.
* Identify metabolic pathways affected and correlate with pregnancy outcomes. 4.6 Research Calculation: 120 participants total (60 per group). 80% power to detect 7% difference in time in range (TIR) between group. Assumptions based on literature, including CONCEPTT study standard deviation 4.7 Ethical Approval: Study will follow Declaration of Helsinki. Institutional ethics approval obtained 5. Research Environment: The study will be conducted at 3-4 major medical centers in Israel with expertise in high-risk pregnancies. Qualified clinical staff including doctors, nurses, dietitians and researchers will be involved in participant recruitment, intervention delivery, data collection and analysis. Necessary equipment like CGMs, metabolomics instruments, etc. are available at these sites.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant women with singleton pregnancies.

  * Over 18 years old.
  * Diagnosis of GDM- 3-h 100-g OGTT according to the American College of Obstetricians and Gynecologists supported by the American Diabetes Association, Or Diagnosis of type 1 or 2 diabetes before pregnancy, Or Diagnosis of early GDM by either OGTT in the first trimester or elevated blood glucose measurements in the fasting (above 95mg/dl) or the postprandial (above 140 mg/dl) state.
  * Are already on or intended to start intensive insulin treatment (at leased 2 injections of insulin per day) or wear an insulin pump.
  * Are willing to wear a continuous glucose monitoring system.
  * BMI of 18.5-42 kg/m2 at the time of diagnosis.

Exclusion Criteria:

* Individual with risk factors for:

  * Placental insufficiency.
  * Hypertension.
  * Renal disease.
  * Thrombophilia
  * Rheumatologic disease.
  * A history of preeclampsia, or fetal growth restriction (IUGR).
  * Individuals with a history of preterm labor, or concomitant therapy with β-blockers or glucocorticoids.
  * Individuals who smoke and/or consume any amount of alcohol during pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Time in range | 24 hours
  Percentage of time during the day that the patient is in the normal range of glucose balance in pregnancy
Time above range | 24 hours
  Percentage of time during the day that the patient is above the normal range of glucose balance in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vounzoulaki E, Khunti K, Abner SC, Tan BK, Davies MJ, Gillies CL. Progression to type 2 diabetes in women with a known history of gestational diabetes: systematic review and meta-analysis. BMJ. 2020 May 13;369:m1361. doi: 10.1136/bmj.m1361. PMID 32404325
- [Background] Petry CJ. Gestational diabetes: risk factors and recent advances in its genetics and treatment. Br J Nutr. 2010 Sep;104(6):775-87. doi: 10.1017/S0007114510001741. Epub 2010 May 21. PMID 20487576
- [Background] McIntyre HD, Catalano P, Zhang C, Desoye G, Mathiesen ER, Damm P. Gestational diabetes mellitus. Nat Rev Dis Primers. 2019 Jul 11;5(1):47. doi: 10.1038/s41572-019-0098-8. PMID 31296866
- [Background] Sweeting A, Wong J, Murphy HR, Ross GP. A Clinical Update on Gestational Diabetes Mellitus. Endocr Rev. 2022 Sep 26;43(5):763-793. doi: 10.1210/endrev/bnac003. PMID 35041752
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Jeffrie Seley J, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 15. Management of Diabetes in Pregnancy: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S254-S266. doi: 10.2337/dc23-S015. PMID 36507645
- [Background] lD Meyers, JP Hellwig JO. Institute of Medicine. Dietary Reference Intakes: The Essential Guide to Nutrient Requirements. 2006.
- [Background] Sweeting A, Mijatovic J, Brinkworth GD, Markovic TP, Ross GP, Brand-Miller J, Hernandez TL. The Carbohydrate Threshold in Pregnancy and Gestational Diabetes: How Low Can We Go? Nutrients. 2021 Jul 28;13(8):2599. doi: 10.3390/nu13082599. PMID 34444759
- [Background] Tanner HL, Ng HT, Murphy G, Barrett HL, Callaway LK, McIntyre HD, Nitert MD. Habitual carbohydrate intake is not correlated with circulating beta-hydroxybutyrate levels in pregnant women with overweight and obesity at 28 weeks' gestation. Diabetologia. 2024 Feb;67(2):346-355. doi: 10.1007/s00125-023-06044-w. Epub 2023 Nov 16. PMID 37971504
- [Background] Mijatovic J, Louie JCY, Buso MEC, Atkinson FS, Ross GP, Markovic TP, Brand-Miller JC. Effects of a modestly lower carbohydrate diet in gestational diabetes: a randomized controlled trial. Am J Clin Nutr. 2020 Aug 1;112(2):284-292. doi: 10.1093/ajcn/nqaa137. PMID 32537643
- [Background] Shalit1 R, Dayan2 N, Yoeli-Ullman2 R, , T. Cukierman-Yaffe1 3; The relationship between low carbohydrate diet and pregnancy outcomes in women with pre_gestational diabetes: a historical prospective study. EASD [Internet]. Barcelona; 2019. Available from: https://www.easd.org/media-centre/home.html#!resources/the-relationship-between-low-carbohydrate-diet-and-pregnancy-outcomes-in-women-with-pre-gestational-diabetes-a-historical-prospective-study
- [Background] Peterson CM, Jovanovic-Peterson L. Percentage of carbohydrate and glycemic response to breakfast, lunch, and dinner in women with gestational diabetes. Diabetes. 1991 Dec;40 Suppl 2:172-4. doi: 10.2337/diab.40.2.s172. PMID 1748252
- [Background] Major CA, Henry MJ, De Veciana M, Morgan MA. The effects of carbohydrate restriction in patients with diet-controlled gestational diabetes. Obstet Gynecol. 1998 Apr;91(4):600-4. doi: 10.1016/s0029-7844(98)00003-9. PMID 9540949